CLINICAL TRIAL: NCT05616260
Title: Acetazolamide for Obstructive Sleep Apnea to Improve Heart Health
Acronym: ACE-Of-HEARTs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Christopher Schmickl, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 804081
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; OSA; CPAP; Acetazolamide
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide; Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide, then Placebo, then optional open-label CPAP-therapy (Experimental): Subjects will start with a 2-week ACETAZOLAMIDE regimen
  * Day 1-13: Acetazolamide 500mg at bedtime at home
  * Day 14: Acetazolamide 500mg at bedtime in the sleep laboratory
  After a wash-out period, subjects will then cross-over to a 2-week PLACEBO regimen:
  * Day 1-13: Placebo (matching Acetazolamide 500mg) at bedtime at home
  * Day 14: Placebo (matching Acetazolamide 500mg) at bedtime in the sleep laboratory
  After a wash-out period, subjects may then undergo an OPTIONAL, OPEN-LABEL 2-week CPAP regimen:
  - Day 1-14: CPAP will be used at home during sleep
  Interventions: Drug: Acetazolamide; Drug: Placebo; Device: Continuous Positive Airway Pressure
- Placebo, then Acetazolamide, then optional open-label CPAP-therapy (Experimental): Subjects will start with a 2-week PLACEBO regimen
  * Day 1-13: Placebo (matching Acetazolamide 500mg) at bedtime at home
  * Day 14: Placebo (matching Acetazolamide 500mg) at bedtime in the sleep laboratory
  After a wash-out period, subjects will then cross-over to a 2-week ACETAZOLAMIDE regimen:
  * Day 1-13: Acetazolamide 500mg at bedtime at home
  * Day 14: Acetazolamide 500mg at bedtime in the sleep laboratory
  After a wash-out period, subjects may then undergo an OPTIONAL, OPEN-LABEL 2-week CPAP regimen:
  - Day 1-14: CPAP will be used at home during sleep
  Interventions: Drug: Acetazolamide; Drug: Placebo; Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide tablet (encapsulated)
  Other Names: Diamox
Drug: Placebo — Sugar capsule manufactured to match encapsulated Acetazolamide
Device: Continuous Positive Airway Pressure — Standard CPAP device
  Other Names: CPAP

SUMMARY:
Obstructive sleep apnea (OSA) is a severe type of snoring causing people to choke in their sleep. It affects millions of Americans, causing many health problems. For example, patients with OSA often feel very sleepy and are at risk of falling asleep while driving. OSA also causes elevated blood pressure increasing the risk for heart attacks and strokes. Patients with OSA are often treated with a face-mask that helps them breath at night but can be difficult to tolerate. In fact, about half the patients eventually stop using this mask. Because there are few other treatments (and no drug therapy), many OSA patients are still untreated. Of note, especially young adults (i.e. 18 to 50 years old) benefit from treating their OSA, but they are also less likely to use the mask.

Acetazolamide (a mild diuretic drug) has been used for over 50 years to treat many different conditions and is well tolerated. Recent data suggest, that acetazolamide may help OSA patients to not choke in their sleep and lower their blood pressure. Especially young adults with OSA are likely to respond well to this drug. Further, its low cost (66¢/day) and once- daily dosing may be particularly attractive for young OSA patients unable or unwilling to wear a mask each night. But previous studies had many limitations and did not focus on young adults. The goal of this study is to test if acetazolamide can improve sleep apnea and cardiovascular health in young adults with OSA (18-50 years old), and how it does that. Thus, we will treat 46 young OSA patients with acetazolamide or placebo for 2 weeks each. The order in which participants receive the drug or placebo will be randomized. At the end of each 2 week period we will assess OSA severity and cardiovascular health. Thus, this study will help assess acetazolamide's potential value for OSA treatment, and may also help to identify patients who are most likely to respond to acetazolamide (including select individuals >50 years of age).

Ultimately, this work promises a drug therapy option for millions of OSA patients who are unable to tolerate current treatments.

DETAILED DESCRIPTION:
The goal of this randomized, controlled, double-blind clinical trial is to compare the medication acetazolamide 500mg/day against placebo in young adults (i.e. 18 to 50 years old) who have obstructive sleep apnea and a high blood pressure. The main questions this trial aims to answer are:

* Is acetazolamide for 2 weeks more effective than placebo for treating obstructive sleep apnea?
* Is acetazolamide for 2 weeks more effective than placebo for improving cardiovascular health including blood pressure?
* What are potential predictors and mechanisms of improvements with acetazolamide in sleep apnea and cardiovascular health?

Participants will undergo the following activities:

* Eligibility screening (online or via phone; ~10min)
* Subjects who screen positive: in-person eligibility assessment (~1h) including a history, exam, blood testing, plus an overnight home sleep test
* Participants who are eligible: will come to the research lab (~15min) and be provided with a 2-week supply of the first study drug (i.e. acetazolamide or placebo) to be taken each night at home. Neither the researchers, nor the participants will know whether participants received acetazolamide or placebo. During this 2-week period, participants will wear a watch-sized activity tracker to measure their sleep amount and researchers will check in on participants weekly; at the end of the 2-week period participants are asked to wear a 24-hour blood pressure monitor and then come in for an overnight visit (~12h) which includes the following activities: general exam, questionnaires, blood test, measures of cardiovascular health (e.g. blood pressure) and neurocognitive function (e.g. a memory test), and an overnight sleep study to assess the severity of sleep apnea
* Participants will then receive a 2-week supply of the other study drug (i.e. acetazolamide or placebo) and repeat all the activities
* Optional: after completing the activities above, participants who are interested in using continuous positive airway pressure (CPAP) and are deemed good candidates for this approach by the investigators, will be offered 2-weeks of CPAP and repeat the same activities as were done when taking the study drugs (except there will be no overnight sleep study).

Researchers will compare the effects of acetazolamide on sleep apnea severity and cardiovascular health with the effects of placebo (and CPAP) to see if acetazolamide may be an effective treatment for select patients with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Body mass index ≤ 35 kg/m2
* Untreated OSA (AHI ≥10/h)
* Abnormal blood pressure (>120/80mmHg, or on stable anti-hypertensive therapy for >1month)

Exclusion Criteria:

* Substantial sleep hypoxemia (SpO2<80% for >10% of the monitoring time during the home sleep test, or for >25% of the total sleep time during any of the in-laboratory studies)
* Severe uncontrolled hypertension (>160/110mmHg during baseline assessment; >180/120mmHg during follow up assessments)
* Abnormally low blood counts/electrolytes or renal function at baseline
* Mean use of OSA therapy ≥ 1h/night during past 1 month, or plans to urgently resume/(re)start clinical OSA therapy within 2 months
* Significant, uncontrolled cardiac, pulmonary, endocrine, renal, hepatic, neurocognitive, psychiatric, or urologic (e.g., kidney stones) disorder
* Other major sleep disorder (e.g., narcolepsy)
* Urgent need to initiate effective OSA therapy (i.e., Epworth sleepiness score >18, commercial driver, prior sleep-related car accident, or based on MD judgment)
* Severe allergy to sulfa-drugs or taking another carbonic-anhydrase inhibitor (e.g., topiramate, zonisamide)
* Pregnancy/breastfeeding (current/planned)
* Prisoners
* Illicit substance abuse or >2 standard drinks of alcohol/day
* Medications that may affect OSA or ventilatory control (e.g., opiates, sedatives)
* Thiazide/loop diuretic (risk of hypokalemia)
* Inability to give consent or follow procedures
* Safety concern based on MD judgment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | 14 days
  The AHI is a measure of sleep apnea severity and is defined as the number of apneas (no breathing for 10+ seconds) and hypopneas (reduced breathing for 10+ seconds associated with a >=3% desaturation or cortical arousal) per hour of sleep.
24-hour Mean Blood Pressure | 14 days
  Based on 24h blood pressure measurements

SECONDARY OUTCOMES:
Hypoxic Burden | 14 days
  Respiratory event-associated area under the desaturation curve from pre-event baseline
Reactive Hyperemia Index | 14 days
  Based on a device called EndoPAT, which measures non-invasively bloodflow before, during, and after 5-minutes of occlusion to one arm.
Response Speed | 14 days
  Based on 10-minute Psychomotor vigilance task (PVT)
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SDA) instrument | 14 days
  Based on response pattern scoring, the PROMIS 8-item SDA score will be converted into a T-score with a mean of 50 (reflecting the average for the United States general population) and a standard deviation of 10. Higher t-scores reflect greater sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment (SRI) instrument | 14 days
  Based on response pattern scoring, the PROMIS 8-item SRI score will be converted into a T-score with a mean of 50 (reflecting the average for the United States general population) and a standard deviation of 10. Higher t-scores reflect greater sleep-related impairment.
Epworth Sleepiness Scale (ESS) | 14 days
  The ESS is an 8-item instrument assessing the likelihood of dozing off in 8 different situations with points for each item ranging from 0 to 3 (0 = would never doze off; 3 = high chance of dozing off). The points for each item are summed up, thus the total score ranges from 0 to 24, with higher ESS scores indicating greater sleepiness.
24-hour Mean Systolic Blood Pressure | 14 days
  Based on 24h blood pressure measurements
24-hour Mean Diastolic Blood Pressure | 14 days
  Based on 24h blood pressure measurements

OTHER OUTCOMES:
Measures of Heart-rate Variability | 14 days
  Based on 5 min awake, supine ECG sampled at >250Hz
Overnight Memory Improvement (%) | 14 days
  Based on Verbal Paired-Associates task
Short Form 36 (SF-36) Health Survey | 14 days
  The SF36 is a widely used questionnaire to measure general health-related quality of life across 8 domains (e.g. physical functioning, Energy/fatigue, Social functioning, etc). The score for each of the 8 domains ranges from 0 to 100, with greater scores indicating better health-related quality fo life in this domain.
Sleep Apnea Traits with special focus on loop gain | 14 days
  Quantified from routine polysomnography data.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Schmickl, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego; Altman Clinical and Translational Research Institute Building, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No